CLINICAL TRIAL: NCT06966921
Title: The Effect of Cranial Electrotherapy Stimulation on the Cognition, Anxiety, Depression and Sleep Quality of Chronic Psychiatric Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liu Hsing Yu (Other)
Responsible Party: Sponsor-Investigator, Liu Hsing Yu, nurse, TsaoTun Psychiatric Center, Department of Health, Taiwan
Organization: TsaoTun Psychiatric Center, Department of Health, Taiwan (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 113019
Record Dates: First submitted 2025-04-17; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Sleep; Depression Disorders
Keywords: Cranial Electrotherapy Stimulation; Chronic Psychiatric Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): the experimental group was provided with 5 CES participations per week, each time for 40 minutes, for a total of 12 weeks
  Interventions: Device: CES
- control group (No Intervention)

INTERVENTIONS:
Device: CES — Currently, most CES intervention studies are applied to the general public, and a few studies focus on athletic performance. There are no related studies on residents of psychiatric nursing homes, nor are there any research designs for improving cognitive impairment. Therefore, this study explores the use of CES programs to improve the cognition, anxiety, depression, and other conditions of residents of psychiatric care homes, with the goal of improving their quality of life.
  Arms: experimental group

SUMMARY:
1. Research background Residents of nursing homes are chronically ill patients who are placed in long-term homes. Studies have shown that most residents live alone and are prone to loneliness, loss, depression, and anxiety (Lapane et al., 2022). Cranial electrostimulation (CES) can improve anxiety, depression, and sleep, but there are few studies on the cognitive status of patients with chronic mental illness.
2. Research purpose This study uses cranial microcurrent stimulation (CES) to improve cognition, anxiety, depression, sleep and other conditions in patients with chronic mental illness, with the aim of improving their quality of life.
3. Screening criteria for respondents 3.1 Inclusion criteria (Those who meet the following criteria are suitable to participate in this study)

1. Chronic mental illness patients, 2. Mini-Mental State Examination (MMSE) ≥ 16 points, 3. Education level is junior high school graduates or above, 4. Appropriate oral expression ability, 5. Those who can complete the research consent form, 6. Those who are willing to participate in this study Exclusion conditions (If you have the following conditions, you cannot participate in this study)

1. Those with obvious risk of violence or suicide; 2. Those with cognitive impairment diagnosed with intellectual disability or autism 4. Research Methods

1. The study was conducted at the Psychiatric Center
2. A total of 92 people were admitted, and they were randomly grouped.
3. This study is a interventional study. Before the intervention, a questionnaire must be filled out, which takes about 30 minutes. Then CES is performed 5 times a week, each time for 40 minutes. After completion, the questionnaire must be filled out again. After 3 months of follow-up, another questionnaire test will be conducted.
4. Possible discomfort and treatment methods During the CES intervention, if you feel dizzy, skin allergies, ear discomfort, or any discomfort, the intervention will be stopped immediately and the medical team will evaluate and treat you.
5. Expected benefits of the study This study uses cranial electrostimulation (CES) to improve cognition, anxiety, depression, sleep and other conditions in patients with chronic mental illness, with the aim of improving their quality of life.

6 Matters that respondents should cooperate with during the research Express your true inner thoughts on the questionnaire content. 7 Confidentiality This study collects data through questionnaires. All identifiable data will be coded to ensure personal data security and case privacy.

8. Subsidies and Damages Respondents who complete the research data collection will receive a gift voucher worth approximately NT$300

ELIGIBILITY:
Inclusion Criteria:

* 1. Chronic mental illness patients, 2. Mini-Mental State Examination (MMSE) ≥ 16 points, 3. Education level is junior high school graduates or above, 4. Appropriate oral expression ability, 5. Those who can complete the research consent form, 6. Those who are willing to participate in this study

Exclusion Criteria:

* 1. Those with obvious risk of violence or suicide 2. People with cognitive impairment who have been diagnosed with mental retardation or autism

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
sleep | "From enrollment to the end of treatment at 12 weeks"
  The Pittsburgh Sleep Quality Inventory (PSQI) is a self-administered questionnaire developed by Buysse et al. (1989). They felt that sleep quality has become an important issue in clinical practice, so they referred to the existing sleep quality scale and developed it into a self-administered questionnaire that can explore sleep conditions in the past month. This scale can be used as a self-assessment tool to measure sleep quality. Its content covers seven sub-concepts, including self-assessed sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbance, use of sleeping pills, and daytime function.
Depression | "From enrollment to the end of treatment at 12weeks"
  This study used the Taiwanese Depression Scale (TDS) revised by scholar Yu (2011). The purpose of this scale is to screen cases with depressive symptoms. It has a total of 18 questions, and each question is divided into 0 points (no or very few symptoms), 1 point (sometimes there are symptoms), 2 points (often there are symptoms), and 3 points (often or always there are symptoms) according to the severity. The total score ranges from 0 to 54 points. The higher the score, the more severe the depressive symptoms (Yu, Huang, and Liu, 2011).
  Lee et al. conducted a reliability and validity analysis on 107 community residents using this scale and found that the internal consistency Cronbach's alpha coefficient was 0.90.
  The DSM III-R (Edition, Revised) was used as the diagnostic standard. After the receiver operating characteristic curve (ROC) analysis, it was found that the total score of 19 points was the best cut-off point for diagnosing depression, with a sensitivity of 0.89 and a speci

SECONDARY OUTCOMES:
cognition | "From enrollment to the end of treatment at 12 weeks"
  In this study, the Chinese version of the Montreal Cognitive Assessment (MoCA) was used to assess the cognitive status of the cases. The test was administered once before and after the intervention to evaluate whether the intervention measures had an effect on improving the cognitive function of the cases.
anxiety | "From enrollment to the end of treatment at 12 weeks"
  This study used the State-Trait Anxiety Inventory to assess the anxiety status of the patients. The test was administered once before and after the intervention to assess whether the intervention measures had an effect on improving the anxiety of the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Tsaotun Psychiatric Center, MOHW, Nantou City, Taiwan

IPD SHARING:
Plan to Share IPD: No